CLINICAL TRIAL: NCT05034328
Title: Impact of Adding Healsea® Isotonic Nasal Spray to Conventional Therapies for the Care of Children With Allergic Rhinitis Presenting With Symptoms of Acute Infectious Rhinitis: an Observational Study
Brief Title: Symbiofilm Trial in Allergic Kids (SYMBIOFILM-TAK)
Status: Completed | Type: Observational
Sponsor: Lallemand Pharma AG (Industry)
Responsible Party: Sponsor
Other Study IDs: LPH-2101
Record Dates: First submitted 2021-09-02; First posted 2021-09-05 (Actual); Results first posted 2025-01-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2023-03

CONDITIONS: Common Cold; Allergy
Keywords: Infectious rhinitis, nasal irrigation, perennial allergy
MeSH Terms: conditions — Common Cold; Hypersensitivity | interventions — Cold Temperature

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healsea® Children: isotonic seawater based nasal spray supplemented with natural Symbiofilm® extract: Children will receive Healsea® Children nasal spray on top of conventional therapies for common cold, as needed.
  Interventions: Device: Healsea® Children; Other: Conventional therapies for common cold
- Conventional therapies: Children will receive conventional therapies for common cold as needed, nasal irrigation excluded
  Interventions: Other: Conventional therapies for common cold

INTERVENTIONS:
Device: Healsea® Children — Children will be administered Healsea Children , one puff (1-2 sec) in each nostril twice a day for 10 days on top of conventional therapies, as needed
  Other Names: Conventional therapies for common cold
  Groups: Healsea® Children: isotonic seawater based nasal spray supplemented with natural Symbiofilm® extract
Other: Conventional therapies for common cold — Children will receive conventional therapies for common cold, nasal irrigation excluded (antipyretics, mucolytics, decongestants, antitussives, systemic and topical corticosteroids, antibiotics)

SUMMARY:
Healsea® Children is a seawater-based nasal spray supplemented with a natural Symbiofilm® extract (0.02%) isolated from marine bacteria. Symbiofilm has antibiofilm activity against various bacterial pathogens involved in respiratory tract infections.Healsea® Children is indicated in the cleaning and moistening of nasal mucosa during common cold and rhinitis for children above 6 years.

This non interventional post-market clinical investigation aimed to confirm the benefit of Healsea® Children in real life setting in children with perennial allergy who are more prone to common cold.

DETAILED DESCRIPTION:
Healsea® Children is a seawater-based nasal spray supplemented with a natural Symbiofilm® extract (0.02%) isolated from marine bacteria. Symbiofilm® is an exopolymeric composition with emulsifying properties, in vitro antibiofilm activity and detachment properties against various bacterial pathogens involved in respiratory tract infections. Symbiofilm® has no bacteriostatic nor bactericidal activities. Healsea® Children is indicated in the cleaning and moistening of nasal mucosa during common cold and rhinitis.

The common cold is an acute viral infection of the upper respiratory tract, involving, to variable degrees, sneezing, nasal congestion and discharge (rhinorrhea), sore throat, cough, low-grade fever, headache, and malaise (1). It can be caused by members of several families of viruses; the most common are rhinoviruses. Acute viral rhinitis is generally self-limiting. In children where the illness is not self-limiting and extends beyond 7-10 days, many agree that a bacterial infection is likely (1). Bacterial over infections and progression to a chronic state are favoured by the formation of biofilms, which facilitate bacterial growth and persistence as well as reducing antibiotic efficacy (2-3).

Allergic diseases may play a particular role in promoting the respiratory infection recurrences (4). The physiological immune response is impaired in allergic subjects and allergic inflammation favours predisposition to respiratory infections. Subjects with allergic disorders may have functional defect of type 1 immune response that is relevant in fighting infections (5-6).

Allergic rhinitis (AR) may affect up to 40% of the paediatric population. Nasal symptoms are caused by exposure to an allergen to which a patient is sensitized.

AR is characterized by typical nasal symptoms and immunoglobulin E (IgE) -mediated inflammation. The allergic inflammatory process releases many cytokines and other proinflammatory proteins. Inflammation caused by nasal allergy leads to obstruction, fluid accumulation and acute disease. If these diseases are unsuccessfully treated, a chronic state of inflammation, obstruction, and infection develops that can cause mucosal damage and, ultimately, chronic disease (7).

For these reasons, the paediatric IgE-dependent allergic population that is more prone to common cold represents a suitable target for Healsea® Children (8-9).

During this prospective post-market clinical investigation, IgE-dependent allergic children with early symptoms of infectious rhinitis will be followed, children being treated with Healsea® Children on top of common cold conventional therapies or with conventional therapies only (excluded nasal irrigation).

Conventional therapies for non-complicated infectious rhinitis are symptomatic but are not without side effects. For example, decongestant use can increase blood pressure, antihistamine intake is associated with drowsiness.

Healsea® Children represents an interesting alternative that can not only improve acute infectious rhinitis symptomatology but could also limit the complication and progression to chronic state.

This non interventional post-market clinical investigation aimed to confirm the benefit of Healsea® Children in a real life setting in children with perennial allergy.

ELIGIBILITY:
Inclusion Criteria:

1. Male/Female subjects ≥6 and ≤10-year-old
2. AsIgE (Allergy specific IgE) ≥ class 2 (RAST) or positive prick test for at least one perennial allergen
3. Acute infectious rhinitis/rhinosinusitis for ≤48h before trial entry
4. Patient presenting with fever ≥ 37.5 °C at screening
5. Symptoms of headache, muscle ache, chilliness, sore throat, blocked nose, runny nose, cough, sneezing with a total score ≤9 (according to a physician-rated symptom score; scale: 0 to 3 [0: no symptom to 3: severe intensity])
6. At least one of these symptoms: sore throat, runny nose or blocked nose (i.e., with a score ≥1)
7. Written consent obtained from parent/legal guardians
8. Written assent obtained from patient

Exclusion Criteria:

1. Known hypersensitivity/allergy to any component of the test device
2. Medical history that is considered by the investigator as a reason for non-inclusion,
3. Severe nasal septum deviation or other condition that could cause nasal obstruction such as the presence of nasal polyps
4. History of nasal or sinus surgery that in the opinion of the investigator may influence symptom scores
5. Antibiotic intake within 2 weeks before screening
6. Systemic corticosteroids within 4 weeks before screening
7. Antihistamines intake for allergy when treatment was started from less than 4 weeks
8. Bacterial lysate intake within 6 months before screening
9. Chronic decongestant use
10. Recent (within the previous 2 days) intake of a common cold medicine that in the opinion of the investigator may influence symptom score at screening (NSAID, nasal decongestants, cough medicines)

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study population comprises children 6 to10 years old with perennial allergy and early symptoms of common cold.
  The recruitment will be competitive in both group, exposed to Healsea® Children or not exposed to Healsea® Children. However, when 100 patients will be recruited in one group, the recruitment will be stopped in this group but will continue in the other group until 100 patients to be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 186 (Actual)
Dates: Start 2022-02-14 (Actual); Primary Completion 2022-11-03 (Actual); Study Completion 2022-11-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrzej EMERYK, MD, PhD, Principal Investigator — University Children Hospital, Lublin, Poland
Locations (10):
- Poland (10):
  - Research Site, Bialystok
  - Research Site, Bydgoszcz
  - Research Site, Dys
  - Research Site, Głowno
  - Research Site, Krakow
  - Research Site, Lublin
  - Research Site, Rzeszów
  - Research Site, Tarnów
  - Research Site, Warsaw
  - Research Site, Łomża

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fokkens WJ, Lund VJ, Hopkins C, Hellings PW, Kern R, Reitsma S, Toppila-Salmi S, Bernal-Sprekelsen M, Mullol J, Alobid I, Terezinha Anselmo-Lima W, Bachert C, Baroody F, von Buchwald C, Cervin A, Cohen N, Constantinidis J, De Gabory L, Desrosiers M, Diamant Z, Douglas RG, Gevaert PH, Hafner A, Harvey RJ, Joos GF, Kalogjera L, Knill A, Kocks JH, Landis BN, Limpens J, Lebeer S, Lourenco O, Meco C, Matricardi PM, O'Mahony L, Philpott CM, Ryan D, Schlosser R, Senior B, Smith TL, Teeling T, Tomazic PV, Wang DY, Wang D, Zhang L, Agius AM, Ahlstrom-Emanuelsson C, Alabri R, Albu S, Alhabash S, Aleksic A, Aloulah M, Al-Qudah M, Alsaleh S, Baban MA, Baudoin T, Balvers T, Battaglia P, Bedoya JD, Beule A, Bofares KM, Braverman I, Brozek-Madry E, Richard B, Callejas C, Carrie S, Caulley L, Chussi D, de Corso E, Coste A, El Hadi U, Elfarouk A, Eloy PH, Farrokhi S, Felisati G, Ferrari MD, Fishchuk R, Grayson W, Goncalves PM, Grdinic B, Grgic V, Hamizan AW, Heinichen JV, Husain S, Ping TI, Ivaska J, Jakimovska F, Jovancevic L, Kakande E, Kamel R, Karpischenko S, Kariyawasam HH, Kawauchi H, Kjeldsen A, Klimek L, Krzeski A, Kopacheva Barsova G, Kim SW, Lal D, Letort JJ, Lopatin A, Mahdjoubi A, Mesbahi A, Netkovski J, Nyenbue Tshipukane D, Obando-Valverde A, Okano M, Onerci M, Ong YK, Orlandi R, Otori N, Ouennoughy K, Ozkan M, Peric A, Plzak J, Prokopakis E, Prepageran N, Psaltis A, Pugin B, Raftopulos M, Rombaux P, Riechelmann H, Sahtout S, Sarafoleanu CC, Searyoh K, Rhee CS, Shi J, Shkoukani M, Shukuryan AK, Sicak M, Smyth D, Sindvongs K, Soklic Kosak T, Stjarne P, Sutikno B, Steinsvag S, Tantilipikorn P, Thanaviratananich S, Tran T, Urbancic J, Valiulius A, Vasquez de Aparicio C, Vicheva D, Virkkula PM, Vicente G, Voegels R, Wagenmann MM, Wardani RS, Welge-Lussen A, Witterick I, Wright E, Zabolotniy D, Zsolt B, Zwetsloot CP. European Position Paper on Rhinosinusitis and Nasal Polyps 2020. Rhinology. 2020 Feb 20;58(Suppl S29):1-464. doi: 10.4193/Rhin20.600. PMID 32077450
- [Background] Yan J, Bassler BL. Surviving as a Community: Antibiotic Tolerance and Persistence in Bacterial Biofilms. Cell Host Microbe. 2019 Jul 10;26(1):15-21. doi: 10.1016/j.chom.2019.06.002. PMID 31295420
- [Background] Rabin N, Zheng Y, Opoku-Temeng C, Du Y, Bonsu E, Sintim HO. Biofilm formation mechanisms and targets for developing antibiofilm agents. Future Med Chem. 2015;7(4):493-512. doi: 10.4155/fmc.15.6. PMID 25875875
- [Background] Varricchio A, La Mantia I, Brunese FP, Ciprandi G. Inflammation, infection, and allergy of upper airways: new insights from national and real-world studies. Ital J Pediatr. 2020 Feb 10;46(1):18. doi: 10.1186/s13052-020-0782-z. PMID 32039733
- [Background] Ciprandi G, Tosca MA, Fasce L. Allergic children have more numerous and severe respiratory infections than non-allergic children. Pediatr Allergy Immunol. 2006 Aug;17(5):389-91. doi: 10.1111/j.1399-3038.2006.00413.x. PMID 16846459
- [Background] Cirillo I, Marseglia G, Klersy C, Ciprandi G. Allergic patients have more numerous and prolonged respiratory infections than nonallergic subjects. Allergy. 2007 Sep;62(9):1087-90. doi: 10.1111/j.1398-9995.2007.01401.x. Epub 2007 Jun 18. PMID 17578494
- [Background] Eifan AO, Durham SR. Pathogenesis of rhinitis. Clin Exp Allergy. 2016 Sep;46(9):1139-51. doi: 10.1111/cea.12780. PMID 27434218
- [Background] De Corso E, Lucidi D, Cantone E, Ottaviano G, Di Cesare T, Seccia V, Paludetti G, Galli J. Clinical Evidence and Biomarkers Linking Allergy and Acute or Chronic Rhinosinusitis in Children: a Systematic Review. Curr Allergy Asthma Rep. 2020 Sep 5;20(11):68. doi: 10.1007/s11882-020-00967-9. PMID 32889648
- [Background] Lin SW, Wang SK, Lu MC, Wang CL, Koo M. Acute rhinosinusitis among pediatric patients with allergic rhinitis: A nationwide, population-based cohort study. PLoS One. 2019 Feb 12;14(2):e0211547. doi: 10.1371/journal.pone.0211547. eCollection 2019. PMID 30753196

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were outpatients visiting a physician in Polish hospitals or private practices at the onset of a common cold. The first patient was screened and enrolled on 14th of February 2022 and the last patient on 20th October 2022.
Period: Overall Study
Arm/Group | Healsea® Children: Isotonic Seawater Based Nasal Spray Supplemented With Natural Symbiofilm® Extract | Conventional Therapies
Started | 101 | 85
Full Analysis Set (FAS) | 101 (All included subjects who used the investigational device at least once) | 85
Per Protocol Set (PP) (Efficacy population based on the Full Analysis Set without patients with major protocol deviation) | 91 | 76
Completed | 100 | 75
Not Completed | 1 | 10
Not completed — Protocol Violation | 1 | 0
Not completed — Lost to Follow-up | 0 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Healsea® Children: Isotonic Seawater Based Nasal Spray Supplemented With Natural Symbiofilm® Extract | Conventional Therapies | Total
Number analyzed (Participants) | 101 | 85 | 186
Age, Continuous [Mean (Standard Deviation); unit: Years] | 7.86 (1.42) | 8.02 (1.40) | 7.93 (1.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 36 | 81
  Male | 56 | 49 | 105
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 101 | 85 | 186
Region of Enrollment [Number; unit: participants]
  Poland | 101 | 85 | 186
Symptoms of acute rhinitis at baseline: temperature [Mean (Standard Deviation); unit: Degrees Celcius] | 37.75 (0.23) | 37.81 (0.39) | 37.78 (0.31)
Symptoms of acute rhinitis at baseline [Mean (Standard Deviation); unit: units on a scale] — Symptoms of headache, muscle ache, chilliness, sore throat, blocked nose, runny nose, cough, sneezing at baseline according to a physician-rated symptom score for each symptom; scale: 0 → 3 [0: no symptom to 3: severe intensity])
  units on a scale
    Headache | 0.6 (0.6) | 0.5 (0.6) | 0.6 (0.6)
    Muscle ache | 0.1 (0.4) | 0.2 (0.5) | 0.2 (0.4)
    Chiliness | 0.2 (0.4) | 0.3 (0.5) | 0.2 (0.5)
    Sore throat | 0.8 (0.7) | 0.8 (0.7) | 0.8 (0.7)
    Blocked nose | 1.7 (0.7) | 1.6 (0.8) | 1.7 (0.7)
    Runny nose | 1.5 (0.7) | 1.5 (0.7) | 1.5 (0.7)
    Cough | 0.9 (0.8) | 1.1 (1.0) | 1.0 (0.9)
    Sneezing | 1.0 (0.7) | 0.9 (0.7) | 1.0 (0.7)

OUTCOME MEASURES:

1. Primary Outcome: AUC (Area Under Curve) of the Wisconsin Upper Respiratory Symptoms Survey for Kids (WURSS-K) During the 10-day Treatment Period
Description: The WURSS-K will be assessed once daily, from Day1 to Day10 (treatment period) WURSS-K is a 3-dimensional structure questionnaire specifically designed for children 4 to 10 years of age.
  It includes 6 items assessing symptoms (symptoms score: runny nose, stuffy nose, sneezing, sore throat, cough, feeling tired), 7 items assessing functional impairments (quality of life score: think, sleep, breathe, talk, walk/climb stairs/exercise, go to school, play with friends), 1 item assessing global severity. All these items are scored from 0 (absent or no impairment) through 1 (a little bad), 2 (bad) and 3 (very bad). The AUC value of the WURSS-K during the 10 day- treatment period is comprised between 0 WURSS-K score*day (no impairement) and 420 WURSS-K score *day (maximal impairement)
Time Frame: Cumulative AUC of the WURSS score assessed from Day 1 to Day 10
Population: All included subjects who used the investigational medical device at least once and with non-missing value at Day1 and at least another non-missing time point between Day2 and Day10. Otherwise, the AUC was missing.
Measure: Mean (Standard Deviation); unit: scores on WURSS-K scale* days
Arm/Group | Healsea® Children: Isotonic Seawater Based Nasal Spray Supplemented With Natural Symbiofilm® Extract | Conventional Therapies
Number analyzed (Participants) | 101 | 85
scores on WURSS-K scale* days | 36.56 (21.14) | 55.54 (27.86)
Statistical Analysis 1: Comparison: Healsea® Children: Isotonic Seawater Based Nasal Spray Supplemented With Natural Symbiofilm® Extract vs Conventional Therapies; Test type: Superiority; p < 0.05, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Number of Days With Runny Nose
Description: During the treatment period, the WURSS-K will be assessed once daily. After D10, the WURSS-K will be assessed once daily until the subject feels not sick for two consecutive days. Items 2 to 7 will be used to assess the duration of each common cold symptoms in both groups. Runny nose is the item 2
Time Frame: Number of days with runny nose during the 10-day treatment period and a follow-up of 20 days, up to 30 days
Population: All included subjects who used the investigational medical device at least once
Measure: Mean (Standard Error); unit: Day
Arm/Group | Healsea® Children: Isotonic Seawater Based Nasal Spray Supplemented With Natural Symbiofilm® Extract | Conventional Therapies
Number analyzed (Participants) | 101 | 85
Day | 7.4 (6.9) | 9.4 (7.9)
Statistical Analysis 1: Comparison: Healsea® Children: Isotonic Seawater Based Nasal Spray Supplemented With Natural Symbiofilm® Extract vs Conventional Therapies; For each item 2 to 7 of the WURSS-K questionnaire, the impact of the treament chosen on the corresponding common cold symptom duration was analyzed by means of Cox model and p-value (Wald) calculated; Test type: Superiority; p = 0.7026, Regression, Cox; Hazard Ratio (HR) = 1.063, 95% CI 2-sided [0.778 to 1.451]

3. Secondary Outcome: Number of Days With Stuffy Nose
Description: During the treatment period, the WURSS-K will be assessed once daily. After D10, the WURSS-K will be assessed once daily until the subject feels not sick for two consecutive days. Items 2 to 7 will be used to assess the duration of each common cold symptoms in both groups. Stuffy nose is the item 3.
Time Frame: Number of days with stuffy nose during the 10-day treatment period and a follow-up period of 20 days, up to 30 days
Population: FAS
Measure: Mean (Standard Error); unit: Day
Arm/Group | Healsea® Children: Isotonic Seawater Based Nasal Spray Supplemented With Natural Symbiofilm® Extract | Conventional Therapies
Number analyzed (Participants) | 101 | 85
Day | 6.8 (6.3) | 8.6 (7.5)
Statistical Analysis 1: Comparison: Healsea® Children: Isotonic Seawater Based Nasal Spray Supplemented With Natural Symbiofilm® Extract vs Conventional Therapies; For each item 2 to 7 of the WURSS-K questionnaire, the impact of the treatment chosen on the corresponding common cold symptom duration was analyzed by means of Cox model and p-value (Wald) calculated; Test type: Superiority; p = 0.6322, Regression, Cox; Hazard Ratio (HR) = 1.078, 95% CI 2-sided [0.792 to 1.469]

4. Secondary Outcome: Number of Days With Sneezing
Description: During the treatment period, the WURSS-K will be assessed once daily. After D10, the WURSS-K will be assessed once daily until the subject feels not sick for two consecutive days. Items 2 to 7 will be used to assess the duration of common cold symptoms in both groups. Sneezing is the item 4.
Time Frame: Number of days with sneezing during the 10-day treatment period and a follow-up of 20 days, up to 30 days
Population: FAS
Measure: Mean (Standard Error); unit: Day
Arm/Group | Healsea® Children: Isotonic Seawater Based Nasal Spray Supplemented With Natural Symbiofilm® Extract | Conventional Therapies
Number analyzed (Participants) | 101 | 85
Day | 6.1 (6.5) | 5.9 (6.0)
Statistical Analysis 1: Comparison: Healsea® Children: Isotonic Seawater Based Nasal Spray Supplemented With Natural Symbiofilm® Extract vs Conventional Therapies; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.9598, Regression, Cox; Hazard Ratio (HR) = 0.992, 95% CI 2-sided [0.726 to 1.356]

5. Secondary Outcome: Number of Days With Sore Throat
Description: During the treatment period, the WURSS-K will be assessed once daily. After D10, the WURSS-K will be assessed once daily until the subject feels not sick for two consecutive days. Items 2 to 7 will be used to assess the duration of each common cold symptoms in both groups. Sore throat is the item 5.
Time Frame: Number of days with sore throat during the 10-day treatment period and a follow-up of 20 days, up to 30 days
Population: FAS
Measure: Mean (Standard Error); unit: Day
Arm/Group | Healsea® Children: Isotonic Seawater Based Nasal Spray Supplemented With Natural Symbiofilm® Extract | Conventional Therapies
Number analyzed (Participants) | 101 | 85
Day | 3.9 (5.6) | 5.2 (6.9)
Statistical Analysis 1: Comparison: Healsea® Children: Isotonic Seawater Based Nasal Spray Supplemented With Natural Symbiofilm® Extract vs Conventional Therapies; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.1016, Regression, Cox; Hazard Ratio (HR) = 1.333, 95% CI 2-sided [0.945 to 1.880]

6. Secondary Outcome: Number of Days With Cough
Description: During the treatment period, the WURSS-K will be assessed once daily. After D10, the WURSS-K will be assessed once daily until the subject feels not sick for two consecutive days. Items 2 to 7 will be used to assess the duration of each common cold symptoms in both groups. Cough is the item 6.
Time Frame: Number of days with cough during the 10-day treatment period and a follow-up of 20 days, up to 30 days
Population: FAS
Measure: Mean (Standard Error); unit: Day
Arm/Group | Healsea® Children: Isotonic Seawater Based Nasal Spray Supplemented With Natural Symbiofilm® Extract | Conventional Therapies
Number analyzed (Participants) | 101 | 85
Day | 6.1 (6.2) | 7.1 (7.2)
Statistical Analysis 1: Comparison: Healsea® Children: Isotonic Seawater Based Nasal Spray Supplemented With Natural Symbiofilm® Extract vs Conventional Therapies; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.3954, Regression, Cox; Hazard Ratio (HR) = 1.153, 95% CI 2-sided [0.830 to 1.601]

7. Secondary Outcome: Number of Days With "Feeling Tired"
Description: During the treatment period, the WURSS-K will be assessed once daily. After D10, the WURSS-K will be assessed once daily until the subject feels not sick for two consecutive days. Items 2 to 7 will be used to assess the duration of each common cold symptoms in both groups. Feeling tired is the item 7.
Time Frame: Number of days with "feeling tired" during the 10-day treatment period and a follow-up of 20 days, up to 30 days
Population: FAS
Measure: Mean (Standard Error); unit: Day
Arm/Group | Healsea® Children: Isotonic Seawater Based Nasal Spray Supplemented With Natural Symbiofilm® Extract | Conventional Therapies
Number analyzed (Participants) | 101 | 85
Day | 4.8 (6.2) | 6.4 (7.3)
Statistical Analysis 1: Comparison: Healsea® Children: Isotonic Seawater Based Nasal Spray Supplemented With Natural Symbiofilm® Extract vs Conventional Therapies; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 1.218, Regression, Cox; Hazard Ratio (HR) = 1.218, 95% CI 2-sided [0.871 to 1.703]

8. Secondary Outcome: Respiratory Complication Requiring Antibiotic Prescription After the10-day Treatment Period
Description: The number of subjects who develop respiratory complication requiring antibiotic prescription during a 20-day follow-up period after the treatment period will be assessed in both groups and compared
Time Frame: Number of subjects with respiratory complications during the 20-day follow-up period
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Conventional Therapies | Healsea® Children: Isotonic Seawater Based Nasal Spray Supplemented With Natural Symbiofilm® Extract
Number analyzed (Participants) | 85 | 101
Participants | 1 | 2
Statistical Analysis 1: Comparison: Conventional Therapies vs Healsea® Children: Isotonic Seawater Based Nasal Spray Supplemented With Natural Symbiofilm® Extract; The impact of the treatment chosen on the risk to develop respiratory complication requiring antibiotic prescription during a 20-day follow-up was analyzed by a multivariate logistic model; Test type: Superiority; p > 0.05, Regression, Logistic

9. Secondary Outcome: Number of Participants With Use of Concomitant Treatments
Description: Number of subjects who took at least one concomitant treatment (antibiotics, antipyretics, systemic or local mucolytics, decongestants, antitussives, systemic and topical corticosteroids) that may impact symptoms of common cold and comparaison between groups
Time Frame: During 10-day treatment period and a follow-up period of 20 days, up to 30 days
Measure: Number; unit: participants
Arm/Group | Healsea® Children: Isotonic Seawater Based Nasal Spray Supplemented With Natural Symbiofilm® Extract | Conventional Therapies
Number analyzed (Participants) | 101 | 85
participants | 53 | 66
Statistical Analysis 1: Comparison: Healsea® Children: Isotonic Seawater Based Nasal Spray Supplemented With Natural Symbiofilm® Extract vs Conventional Therapies; Test type: Superiority; p = 0.0010, Regression, Logistic; Odds Ratio (OR) = 0.335, 95% CI 2-sided [0.174 to 0.644]

ADVERSE EVENTS:
Time Frame: Adverse events were collected during a 10-day treatment period and a follow-up period of 20 days, up to 30 days
Arm/Group | Healsea® Children: Isotonic Seawater Based Nasal Spray Supplemented With Natural Symbiofilm® Extract | Conventional Therapies
All-Cause Mortality (participants affected / at risk) | 0/101 | 0/85
Serious Adverse Events (participants affected / at risk) | 0/101 | 0/85
Other Adverse Events (participants affected / at risk) | 17/101 | 23/85
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Healsea® Children: Isotonic Seawater Based Nasal Spray Supplemented With Natural Symbiofilm® Extract (N=101) | Conventional Therapies (N=85)
cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 11 (11)
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pharyngitis (Infections and infestations) | 2 (2) | 4 (4)
Bronchitis (Infections and infestations) | 1 (1) | 2 (2)
Rhinitis (Infections and infestations) | 1 (1) | 2 (2)
conjunctivitis (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Tonsilitis (Infections and infestations) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 5 (5) | 3 (3)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 3 (3)
Headache (Nervous system disorders) | 1 (1) | 2 (4)

LIMITATIONS AND CAVEATS:
This is a not blinded, nor placebo-controlled investigation

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2021-09-08): https://cdn.clinicaltrials.gov/large-docs/28/NCT05034328/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-26): https://cdn.clinicaltrials.gov/large-docs/28/NCT05034328/SAP_001.pdf